CLINICAL TRIAL: NCT03075878
Title: A Phase 1B/2, Multicenter, Open-Label, Safety, Tolerability, and Activity Study of SYNT001 in Patients With Warm Autoimmune Hemolytic Anemia (WAIHA)
Brief Title: A Safety Study of SYNT001 in Participants With Warm Autoimmune Hemolytic Anemia (WAIHA)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Focus resources on a planned phase 2/3 study
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SYNT001-102
Record Dates: First submitted 2017-03-03; First posted 2017-03-09 (Actual); Results first posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Warm Autoimmune Hemolytic Anemia
MeSH Terms: interventions — orilanolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: ALXN1830 (Experimental): SYNT001 Dose 1
  Interventions: Drug: ALXN1830
- Cohort 2: ALXN1830 (Experimental): SYNT001 Dose 2
  Interventions: Drug: ALXN1830

INTERVENTIONS:
Drug: ALXN1830 — Administered via IV infusion.
  Other Names: SYNT001

SUMMARY:
This main study objective was to evaluate the safety and tolerability of intravenous (IV) SYNT001 (ALXN1830) in participants with WAIHA.

DETAILED DESCRIPTION:
This study planned to evaluate 2 cohorts: Cohort 1, up to 8 participants to receive IV doses of ALXN1830 (SYNT001 Dose 1); Cohort 2, up to 12 participants to receive IV doses of ALXN1830 (SYNT001 Dose 2).

This study was terminated after the safety, tolerability, pharmacokinetics, pharmacodynamics, and efficacy were characterized in participants with WAIHA in Cohort 1 (SYNT001 Dose 1), before any participants were enrolled in Cohort 2.

ELIGIBILITY:
Inclusion Criteria:

Participants had to meet the following criteria to be included:

* Willing and able to read, understand, and sign an informed consent form
* Confirmed diagnosis of WAIHA by enrolling physician
* Must have used medically acceptable contraception

Exclusion Criteria:

Participants who met any of the following criteria were excluded:

* Participant unable or unwilling to comply with the protocol
* Active non-hematologic malignancy or history of non-hematologic malignancy in the 3 years prior to screening (exclusive of non-melanoma skin cancer and cervical cancer in situ)
* Positive for human immunodeficiency virus or hepatitis C antibody
* Positive for hepatitis B surface antigen
* Any exposure to an investigational drug or device within the 30 days prior to screening
* Intravenous immunoglobulin treatment within 30 days of screening
* Plasmapheresis or immunoadsorption within 30 days of screening
* Participant had any current medical condition that, in the opinion of the Investigator, may have compromised their safety or compliance, precluded successful conduct of the study, or interfered with interpretation of the results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-08-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (9):
  - Alexion Study Site, Los Angeles, California
  - Alexion Study Site, San Francisco, California
  - Alexion Study Site, Boston, Massachusetts
  - Alexion Study Site, Pittsfield, Massachusetts
  - Alexion Study Site, Rochester, Minnesota
  - Alexion Study Site, Cleveland, Ohio
  - Alexion Study Site, Philadelphia, Pennsylvania
  - Alexion Study Site, Pittsburgh, Pennsylvania
  - Alexion Study Site, Seattle, Washington
- Alexion Study Site, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was terminated after the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and efficacy were characterized in Cohort 1 (SYNT001 Dose 1), before any participants were enrolled in Cohort 2 (SYNT001 Dose 2). This results disclosure is for Cohort 1 only.
Groups:
- Cohort 1: ALXN1830: SYNT001 Dose 1: Participants received ALXN1830.
Period: Overall Study
Arm/Group | Cohort 1: ALXN1830
Started | 8
Received at Least 1 Dose of Study Drug (Safety Population) | 8
Completed | 7
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Safety Population: All participants who received at least 1 dose of study drug.
Arm/Group | Cohort 1: ALXN1830
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (16.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Age at Warm Autoimmune Hemolytic Anemia Diagnosis [Mean (Standard Deviation); unit: years] | 48.4 (16.85)

OUTCOME MEASURES:

1. Primary Outcome: Count Of Participants Reporting Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE was defined as any adverse event that starts on or after the first dose of study drug or occurs prior to the first dose and worsens in severity on or after the first dose of study drug, during the Treatment Period and Follow-up Period. A TEAE was considered "serious" if, in the view of either the investigator or sponsor, it resulted in any of the following outcomes: death, life-threatening adverse drug event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, congenital anomaly/birth defect, or an event that may have jeopardized the participant and may have required medical or surgical intervention to prevent one of the previously listed outcomes. A summary of serious and all other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module. All serious TEAEs were not considered related to the study drug.
Time Frame: Day 0 (after first dose) through Day 112
Population: Safety Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ALXN1830
Number analyzed (Participants) | 8
Participants
  TEAEs | 8
  Serious TEAEs | 2
  Discontinuations due to TEAEs | 0
  Deaths | 0

2. Secondary Outcome: Maximum Serum Concentration (Cmax) On Day 0 And Day 28
Description: The Cmax was determined directly from the concentration-time profile. Starting on Days 0 and 28, serum samples were collected just prior to the start of study drug infusion (predose), at 5 minutes, at 2, 4, 6, 24, and 48 hours, and at 5 days postdose after the end-of-study drug infusion. Results are reported in micrograms/milliliter (ug/mL).
Time Frame: Predose, 5 minutes, 2, 4, 6, 24, and 48 hours, and 5 days postdose
Population: PK Population: All participants who received at least 1 dose of study drug and had postdose PK data available at the specified timepoint.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Cohort 1: ALXN1830
Number analyzed (Participants) | 8
ug/mL
  Day 0 | 249.6 (35.76)
  Day 28 | 245.8 (41.55)

3. Secondary Outcome: Change From Baseline In Reticulocyte Count At Day 33
Description: Reticulocyte count was measured as a PD biomarker. Pharmacodynamic samples were collected for analyses throughout the study prior to infusion of study drug for Cohort 1. Measurements for PD biomarkers were derived from the laboratory results. Results are reported in cells/liter (cells*10^12/L). A decrease in reticulocyte count indicated a potential improvement in condition.
Time Frame: Baseline, Day 33
Population: PD Population: All participants who received at least 1 dose of study drug and had postdose PD data available at the specified timepoint.
Measure: Mean (Standard Deviation); unit: cells*10^12/L
Arm/Group | Cohort 1: ALXN1830
Number analyzed (Participants) | 7
cells*10^12/L | -0.044 (0.0948)

4. Secondary Outcome: Change From Baseline In Hemoglobin At Day 33
Description: Hemoglobin was measured as a PD biomarker. Pharmacodynamic samples were collected for analyses throughout the study prior to infusion of study drug for Cohort 1. Measurements for PD biomarkers were derived from the laboratory results. Results are reported in grams/deciliter (g/dL). An increase in hemoglobin indicated a potential improvement in condition.
Time Frame: Baseline, Day 33
Population: PD Population: All participants who received at least 1dose of study drug and had postdose PD data available at the specified timepoint.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Cohort 1: ALXN1830
Number analyzed (Participants) | 8
g/dL | 0.66 (1.581)

5. Secondary Outcome: Immunogenicity Of ALXN1830 At Day 112, As Assessed By Anti-ALXN1830 Antibody Level
Description: Immunogenicity analyses are reported for Day 112. Testing was carried out to detect binding antidrug antibodies by anti-ALXN1830 antibody level. Results are reported as the reciprocal of the titer where they cross the study cut point.
Time Frame: Day 112
Population: Safety Population: All participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: reciprocal of the titer
Arm/Group | Cohort 1: ALXN1830
Number analyzed (Participants) | 4
reciprocal of the titer | 99.220 (165.8149)

ADVERSE EVENTS:
Time Frame: Baseline through Day 112
Arm/Group | Cohort 1: ALXN1830
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 2/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: ALXN1830 (N=8)
Anaemia (Blood and lymphatic system disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: ALXN1830 (N=8)
Fatigue (General disorders) | 2
Chills (General disorders) | 1
Face oedema (General disorders) | 1
Influenza like illness (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Headache (Nervous system disorders) | 4
Dizziness (Nervous system disorders) | 2
Dizziness postural (Nervous system disorders) | 1
Hypersomnia (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Fall (Injury, poisoning and procedural complications) | 1
Infusion-related reaction (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Blepharospasm (Eye disorders) | 1
Haematocrit decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Increased appetite (Metabolism and nutrition disorders) | 1
Restlessness (Psychiatric disorders) | 1
Flushing (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
The study was terminated after the safety, tolerability, PK, PD, and efficacy were characterized in the Warm Autoimmune Hemolytic Anemia participants in Cohort 1 (SYNT001 Dose 1).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can review results communications at least 60 days prior to public release. Within 30 days of receipt, Sponsor shall advise of any information which is Confidential Information (other than Study Data) or which may impair the availability of patent protection for Inventions. Sponsor can require removal of specifically identified Confidential Information (other than Study Data) and/or delay the communication an additional 60 days to enable Sponsor to seek patent protection for Inventions.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/78/NCT03075878/SAP_000.pdf
  • Study Protocol (2018-10-23): https://cdn.clinicaltrials.gov/large-docs/78/NCT03075878/Prot_001.pdf